CLINICAL TRIAL: NCT01612767
Title: The Treatment of Coronary Artery Lesions Using the PRO-Kinetic Energy Cobalt-Chromium, Bare-Metal Stent
Brief Title: BIOHELIX-I Bare Metal Stent Study
Acronym: BIOHELIX-I
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G110147
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Coronary Arteries Disease
Keywords: de novo coronary lesions; restenotic coronary lesions; coronary arteries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pro-Kinetic Energy Stent (Experimental)
  Interventions: Device: PRO-Kinetic Energy Stent

INTERVENTIONS:
Device: PRO-Kinetic Energy Stent — Coronary artery stent implant

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of the investigational BIOTRONIK PRO-Kinetic Energy stent in subjects with atherosclerotic disease of native coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

For a subject to be enrolled in the study and considered for the index procedure, the following initial inclusion criteria must be met:

* Age ≥ 18 years
* Willingness to comply with study follow-up requirements
* Candidate for a percutaneous coronary intervention (PCI) procedure
* Candidate for coronary artery bypass graft surgery
* Documented evidence of stable or unstable angina pectoris or positive functional ischemia study (e.g. exercise treadmill test, thallium stress test, SPECT, stress echocardiogram or cardiac CT) Stable angina pectoris is defined as a documented Canadian Cardiovascular Society Classification of I, II, III or IV Unstable angina pectoris is defined as a documented Braunwald Classification of B & C, I, II, III
* Written informed consent

For a subject to receive an investigational stent, the following procedure-related criteria must be met:

* De novo or restenotic lesion in a native coronary artery; restenotic lesions must have been previously treated with only standard percutaneous transluminal coronary angioplasty (PTCA) (treatment must be > 12 months prior to the index procedure)
* Target lesion must be in a major coronary artery (target vessel). The target vessel includes the entire territory of the left anterior descending artery, left circumflex artery or right coronary artery and any major side branch of the artery.
* A maximum of one target lesion and one non-target lesion may be treated per subject. The lesions must be located in separate coronary arteries, with treatment of the non-target lesion occurring first using commercially available therapy (with exception of brachytherapy).
* Lesions may be one solid lesion or a series of multiple, smaller lesions to be treated as one lesion
* Target lesion must be treatable with a single investigational stent; an additional stent may be used when treating a vessel dissection or another similar intra-procedure complication (use of investigational stent preferred)
* Angiographic evidence of ≥ 50% and < 100% stenosis (by operator visual estimate) with a TIMI flow > 1
* Target lesion length of ≤ 31 mm by operator visual estimate
* Target vessel reference diameter of 2.25 mm to 4.0 mm by operator visual estimate

Exclusion Criteria:

For a subject to be enrolled in the study and considered for the index procedure, the following initial exclusion criteria must not be present:

* Baseline LVEF of < 30%; LVEF may be measured and assessed by standard-of-care echocardiography procedures within 90 days of the index procedure or by a left ventriculogram prior to the index procedure (operator visual assessment).
* PCI in any vessel 30 days prior to the index procedure or planned for within 30 days after the index procedure
* Stroke or transient ischemic attack within the last 6 months prior to enrollment
* Intolerance to contrast agents that cannot be medically managed and/or intolerance to antiplatelet, anticoagulant or thrombolytic medications
* Refusal of blood transfusions
* Any other medical condition, that in the opinion of the investigator, poses an unacceptable risk for implant of a stent according to the study indications
* Pregnant, planning to become pregnant or nursing during the course of the study. Women of child-bearing potential must have a negative blood pregnancy (beta hCG) test. Female subjects who are surgically sterile or post-menopausal are exempt from having a pregnancy test.
* Known allergy to L-605 CoCr alloy (cobalt, chromium, tungsten and nickel) or amorphous silicon carbide
* Life expectancy of less than one year
* Participation in any other clinical investigational device or drug study.
* Subjects may be concurrently enrolled in a post-market study, as long as the post-market study device, drug or protocol does not interfere with the investigational treatment or protocol of this study.

For a subject to receive an investigational stent the following procedure-related criteria must not be present:

* Documented diagnosis of an acute MI within 72 hours of the index procedure and an elevation of Troponin or creatine kinase-MB (CKMB) above the URL (CKMB measurement is not required if CK is normal) at the time of the index procedure (99th percentile of the individual investigative site's normal reference population)

  * For subjects with stable angina and elevated Troponin, CKMB <99% URL is required
* ECG changes consistent with an acute MI within 72 hours of the index procedure. ECG changes consistent with an acute MI include:

> 1 mm ST segment elevation or depression in consecutive leads New left bundle branch block (LBBB) Development of pathological Q-waves in two contiguous leads of the electrocardiogram (ECG)

* Acute coronary syndrome with baseline Troponin > 99% URL
* INR ≥ 1.6
* Concomitant renal failure with serum creatinine level > 2.5 mg/dL
* Unresolved neutropenia (white blood cell count < 3,000 / µL), thrombocytopenia (platelet count < 100,000 / µL) or thrombocytosis (platelet count > 700,000 / µL)
* Unprotected left main coronary artery disease (CAD) (> 50% diameter stenosis by operator visual estimate)
* Target vessel has been treated with any PCI procedure (e.g. PTCA, stent, cutting balloon, atherectomy, etc.) within 12 months prior to the index procedure
* Target lesion has been treated with a stent, cutting balloon or atherectomy any time prior to the index procedure or has been treated with PTCA within 12 months prior to the index procedure
* Target vessel treated with brachytherapy anytime prior to index procedure
* Planned PCI in the target vessel within 9 months after the index procedure
* Target vessel has a non-target lesion with a > 50% stenosis that requires treatment during the index procedure
* Lesions preventing distal perfusion (TIMI flow 0 and 1) prior to wire crossing
* Target lesion is in the left main coronary artery or within 2 mm of the origin of the left anterior descending artery or left circumflex artery by operator visual estimate
* Target lesion is located within a saphenous vein graft or arterial graft
* Target lesion involves a bifurcation - lesion is located in a major coronary artery and involves a side branch with a diameter > 2 mm (by operator visual estimate)
* Presence of a complication following pre-dilatation of target lesion
* Presence of a complication following treatment of a non-target lesion (if applicable)
* Presence of a target vessel/lesion that has excessive tortuousity/angulation or is severely calcified preventing complete inflation of an angioplasty balloon
* Angiographic evidence of thrombus within the target lesion
* Target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion
* Use of cutting balloons, atherectomy or ablative devices immediately prior to investigational stent placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2012-11; Primary Completion 2015-09 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Gupta, MD, Principal Investigator — Oregon Health and Science University
Locations (34):
- United States (27):
  - Phoenix, Arizona
  - Concord, California
  - Mission Viejo, California
  - Danbury, Connecticut
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Gainesville, Georgia
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Lafayette, Louisiana
  - Lewiston, Maine
  - Takoma Park, Maryland
  - Kansas City, Missouri
  - Springfield, Missouri
  - Newark, New Jersey
  - New York, New York
  - Poughkeepsie, New York
  - Gastonia, North Carolina
  - High Point, North Carolina
  - Columbus, Ohio
  - Portland, Oregon
  - Anderson, South Carolina
  - Greenville, South Carolina
  - Amarillo, Texas
  - McKinney, Texas
  - Tyler, Texas
  - Mechanicsville, Virginia
- Medellín, Colombia
- Germany (3):
  - Bad Segeberg
  - Essen
  - Ludwigshafen
- Riga, Latvia
- Netherlands (2):
  - Amsterdam
  - Eindhoven

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pro-Kinetic Energy Stent
Started | 329
Completed | 287
Not Completed | 42

BASELINE CHARACTERISTICS:
Arm/Group | Pro-Kinetic Energy Stent
Number analyzed (Participants) | 329
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 226
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 306
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 305
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  United States | 215
  Germany | 88
  Netherlands | 17
  Latvia | 8
  Colombia | 1
Medical History [Number; unit: Participants]
  Diabetes | 94
  Hypertension | 276
  Hyperlipidemia | 240
  Current smoker | 60
  Smoked within last 5 years | 31
  Never smoked or not within last 5 years | 238
  History of myocardial infarction (MI) | 67
  Prior coronary artery bypass graft (CABG) | 27
  Prior percutaneous coronary revascularization | 100
  Renal insufficiency | 8
Concomitant Medications [Number; unit: Participants]
  Dual Antiplatelet Therapy (DAPT) | 96
  Aspirin | 260
  Antiplatelet - Clopidogrel | 79
  Antiplatelet - Prasugrel | 9
  Antiplatelet - Ticagrelor | 15
  Antiotensin-converting-enzyme (ACE) inhibitor | 135
  Angiotensin II receptor blocker | 78
  Beta blocker | 203
  Statins | 213
  Insulin | 37
  Anti-coagulant | 32
Lesion Location [Number; unit: Participants]
  Left Anterior Descending (LAD) | 122
  Circumflex | 82
  Right | 125
Lesion Length [Mean (Standard Deviation); unit: mm] | 13.7 (6.0)
Vessel Diameter [Mean (Standard Deviation); unit: mm] — MLD = minimal luminal diameter
  mm
    Pre-deployment target vessel MLD | 0.9 (0.4)
    Pre-deployment target vessel reference diameter | 2.9 (0.5)
    Post-deployment target vessel MLD | 3.1 (0.5)
Lesion Calcification [Number; unit: Participants]
  None | 245
  Moderate | 58
  Severe | 26
Thrombolysis in Myocardial Infarction (TIMI) Flow [Number; unit: Participants] — TIMI Flow is a system developed during Thrombolysis in Myocardial Infarction (TIMI) trials for grading severity of stenosis and extent of blood flow through coronary arteries; TIMI grade 0 = no perfusion; grade 1 = penetration with minimal perfusion; grade 2 = partial perfusion; grade 3 = complete perfusion. Grade 0 represents no flow beyond an occlusion, while grade 3 represents normal flow.
  Participants
    0 | 1
    1 | 6
    2 | 24
    3 | 298

OUTCOME MEASURES:

1. Primary Outcome: Target Vessel Failure Rate
Description: The primary endpoint for the Pro-Kinetic Energy Stent is the target vessel failure rate at 9-months post-index procedure. Target vessel failure is defined as cardiac death, myocardial infarction and ischemia-driven target vessel revascularization.
Time Frame: 9 months post-index procedure
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pro-Kinetic Energy Stent
Number analyzed (Participants) | 320
Percentage of participants
  Overall Target Vessel Failure Rate | 9.06 [6.15 to 12.76]
  Cardiac death | 0.95 [0.20 to 2.74]
  Myocardial infarction | 1.58 [0.52 to 3.65]
  Ischemia-driven target vessel revascularization | 7.26 [4.65 to 10.69]

2. Secondary Outcome: Target Vessel Failure Rate
Description: Evaluate the target vessel failure rate at 1, 12, 24, and 36 months post-index procedure. Target vessel failure is defined as cardiac death, myocardial infarction (MI) and ischemia-driven target vessel revascularization.
Time Frame: 1, 12, 24 and 36 months post-index procedure
Population: Long term follow-up data collection is ongoing for the 12, 24 and 36 month intervals.
Measure: Number; unit: Percentage of participants
Arm/Group | PRO-Kinetic Energy Stent
Number analyzed (Participants) | 327
Percentage of participants
  1 Month | 1.22
  12 Months: number analyzed (Participants) | 316
  12 Months | 10.76
  24 Months: number analyzed (Participants) | 309
  24 Months | 13.26
  36 Months: number analyzed (Participants) | 301
  36 Months | 17.61

3. Secondary Outcome: Target Vessel Failure Rate - Contribution of Individual Event Types
Description: Contribution of each event type (cardiac death, myocardial infarction (MI) and ischemia-driven target vessel revascularization) to composite rate of target vessel failure.
Time Frame: 1, 12, 24 and 36 months post-index procedure
Population: Long term follow-up data collection is ongoing for the 12, 24 and 36 month intervals.
Measure: Number; unit: Percentage of participants
Groups:
- PRO-Kinetic Energy Stent - 1 Month; PRO-Kinetic Energy Stent - 12 Months; PRO-Kinetic Energy Stent - 24 Months; PRO-Kinetic Energy Stent - 36 Months: PRO-Kinetic Energy Stent: Coronary artery stent implant
Arm/Group | PRO-Kinetic Energy Stent - 1 Month | PRO-Kinetic Energy Stent - 12 Months | PRO-Kinetic Energy Stent - 24 Months | PRO-Kinetic Energy Stent - 36 Months
Number analyzed (Participants) | 327 | 316 | 309 | 301
Percentage of participants
  Cardiac death | 0.00 | 0.96 | 2.30 | 4.07
  Myocardial infarction | 0.61 | 1.61 | 2.00 | 3.50
  Ischemia-driven target vessel revascularization | 0.61 | 8.97 | 10.23 | 12.46

4. Secondary Outcome: Overall Target Vessel Revascularization Rate
Description: Evaluate the overall target vessel revascularization rate of the PRO-Kinetic Energy stent. The rate includes both ischemia-driven revascularization procedures of the target vessel, as well as revascularization procedures of the target vessel without prior clinical symptoms.
Time Frame: 1, 9, 12, 24 and 36 months post-index procedure
Population: Long term follow-up data collection is ongoing for the 12, 24 and 36 month intervals.
Measure: Number; unit: Percentage of participants
Groups:
- PRO-Kinetic Energy Stent - 9 Month; PRO-Kinetic Energy Stent - 12 Month; PRO-Kinetic Energy Stent - 24 Month; PRO-Kinetic Energy Stent - 36 Month: PRO-Kinetic Energy Stent: Coronary artery stent implant
Arm/Group | Pro-Kinetic Energy Stent - 1 Month | PRO-Kinetic Energy Stent - 9 Month | PRO-Kinetic Energy Stent - 12 Month | PRO-Kinetic Energy Stent - 24 Month | PRO-Kinetic Energy Stent - 36 Month
Number analyzed (Participants) | 327 | 318 | 312 | 303 | 289
Percentage of participants | 0.61 | 7.86 | 9.62 | 11.55 | 13.84

5. Secondary Outcome: Overall Target Lesion Failure Rate
Description: Evaluate the target lesion failure rate of the PRO-Kinetic Energy stent. Target lesion failure includes cardiac death, MI, and ischemia-driven target lesion revascularization.
Time Frame: 1, 9, 12, 24 and 36 months post-index procedure
Population: Long term follow-up data collection is ongoing for the 12, 24 and 36 month intervals.
Measure: Number; unit: Percentage of participants
Arm/Group | Pro-Kinetic Energy Stent - 1 Month | PRO-Kinetic Energy Stent - 9 Month | PRO-Kinetic Energy Stent - 12 Month | PRO-Kinetic Energy Stent - 24 Month | PRO-Kinetic Energy Stent - 36 Month
Number analyzed (Participants) | 327 | 321 | 315 | 308 | 300
Percentage of participants | 1.22 | 8.41 | 9.84 | 11.68 | 15.33

6. Secondary Outcome: Target Lesion Failure Rate - Contribution of Individual Event Types
Description: The contribution of each individual event of cardiac death, myocardial infarction, and ischemia-driven target lesion revascularization to the overall rate of target lesion failure.
Time Frame: 1, 9, 12, 24, and 36 months post-index procedure
Population: Long term follow-up data collection is ongoing for the 12, 24 and 36 month intervals.
Measure: Number; unit: Percentage of participants
Arm/Group | Pro-Kinetic Energy Stent - 1 Month | PRO-Kinetic Energy Stent - 9 Month | Pro-Kinetic Energy Stent - 12 Month | Pro-Kinetic Energy Stent - 24 Month | Pro-Kinetic Energy Stent - 36 Month
Number analyzed (Participants) | 327 | 321 | 315 | 308 | 300
Percentage of participants
  Cardiac death | 0.00 | 0.95 | 0.96 | 2.30 | 4.07
  Myocardial infarction | 0.61 | 1.58 | 1.61 | 2.00 | 3.50
  Ischemia-driven target vessel revascularization | 0.61 | 6.60 | 8.04 | 8.61 | 10.07

7. Secondary Outcome: Overall Target Lesion Revascularization Rate
Description: Evaluate the overall target lesion revascularization rate associated with the PRO-Kinetic Energy stent. The overall target lesion revascularization rate includes both ischemia-driven revascularization procedures of the target lesion, as well as revascularization procedures of the target lesion without prior clinical symptoms.
Time Frame: 1, 9, 12, 24 and 36 months post-index procedure
Population: Long term follow-up data collection is ongoing for the 12, 24 and 36 month intervals.
Measure: Number; unit: Percentage of participants
Groups:
- PRO-Kinetic Energy Stent -24 Month; PRO-Kinetic Energy Stent - 36 Month: PRO-Kinetic Energy Stent: Coronary artery stent implant
Arm/Group | Pro-Kinetic Energy Stent - 1 Month | PRO-Kinetic Energy Stent - 9 Month | PRO-Kinetic Energy Stent - 12 Month | PRO-Kinetic Energy Stent -24 Month | PRO-Kinetic Energy Stent - 36 Month
Number analyzed (Participants) | 327 | 318 | 312 | 303 | 289
Percentage of participants | 0.61 | 7.23 | 8.65 | 9.24 | 10.37

8. Secondary Outcome: Composite of All-cause Mortality and All-cause MI
Description: Characterize the overall safety of the PRO-Kinetic Energy stent by evaluating the composite rate of all-cause mortality and all-cause myocardial infarction.
Time Frame: 1, 9, 12, 24, and 36 months post-index procedure
Population: Long term follow-up data collection is ongoing for the 12, 24 and 36 month intervals.
Measure: Number; unit: Percentage of participants
Arm/Group | Pro-Kinetic Energy Stent - 1 Month | PRO-Kinetic Energy Stent - 9 Month | PRO-Kinetic Energy Stent - 12 Month | PRO-Kinetic Energy Stent - 24 Month | PRO-Kinetic Energy Stent - 36 Month
Number analyzed (Participants) | 326 | 321 | 317 | 314 | 311
Percentage of participants | 0.61 | 3.12 | 3.79 | 7.32 | 11.25

9. Secondary Outcome: All-cause Mortality and All-cause MI - Contribution of Individual Rates
Description: Contribution of the individual rates of mortality and myocardial infarction to the overall composite safety rate.
Time Frame: 1, 9, 12, 24, and 36 months post-index procedure
Population: Long term follow-up data collection is ongoing for the 12, 24 and 36 month intervals.
Measure: Number; unit: Percentage of participants
Arm/Group | Pro-Kinetic Energy Stent - 1 Month | PRO-Kinetic Energy Stent - 9 Month | PRO-Kinetic Energy Stent - 12 Month | PRO-Kinetic Energy Stent - 24 Month | PRO-Kinetic Energy Stent - 36 Month
Number analyzed (Participants) | 326 | 321 | 317 | 314 | 311
Percentage of participants
  All-cause mortality | 0.00 | 1.87 | 2.52 | 5.73 | 8.68
  Cardiac mortality | 0.00 | 0.93 | 0.95 | 2.23 | 3.86
  Non-cardiac mortality | 0.00 | 0.93 | 1.58 | 3.50 | 4.82
  All-cause MI | 0.61 | 1.56 | 1.58 | 1.91 | 3.22

10. Secondary Outcome: Stent Thrombosis Rate
Description: Evaluate the stent thrombosis rate associated with the PRO-Kinetic Energy stent. Stent thrombosis was classified according to both timing and evidence as outlined by the ARC definition of stent thrombosis. Participants were included in the evaluations at visit intervals if they had a visit at the specified interval or a thrombosis was reported at or before the visit.
Time Frame: 1, 9, 12, 24 and 36 months post-index procedure
Population: Long term follow-up data collection is ongoing for the 12, 24 and 36 month intervals.
Measure: Number; unit: Percentage of participants
Arm/Group | Pro-Kinetic Energy Stent - 1 Month | PRO-Kinetic Energy Stent - 9 Month | PRO-Kinetic Energy Stent - 12 Month | PRO-Kinetic Energy Stent - 24 Month | PRO-Kinetic Energy Stent - 36 Month
Number analyzed (Participants) | 327 | 319 | 313 | 305 | 293
Percentage of participants
  Definite stent thrombosis | 0.3 | 0.9 | 1.0 | 1.0 | 1.4
  Probable stent thrombosis | 0.0 | 0.3 | 0.3 | 0.3 | 0.3
  Total definite / probable stent thrombosis | 0.3 | 1.3 | 1.3 | 1.3 | 1.7
  Possible stent thrombosis | 0.0 | 0.9 | 1.0 | 1.6 | 2.7

11. Secondary Outcome: Index Procedure Success
Description: Evaluate the index procedure success associated with the implant of the PR-Kinetic Energy stent. procedure success is defined as the successful delivery and deployment of the investiational stent at the intended target lesion in combination with any adjunctive device (if applicable) to attain a final residual stenosis of < 30% by operator visual estimate without the occurrence of cardiac death, any MI (target vessel or non-target vessel) or TLR prior to hospital discharge.
Time Frame: Index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Pro-Kinetic Energy Stent
Number analyzed (Participants) | 329
Percentage of participants | 98.8

12. Secondary Outcome: Device Success During the Index Procedure
Description: Evaluate the device success associated with the implant of the PRO-Kinetic Energy stent. Device success is defined as the successful delivery and deployment of the investigational stent at the intended target lesion in combination with standard post-dilation (if applicable) to attain a final residual stenosis of < 30% by operator visual estimate.
Time Frame: Index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Pro-Kinetic Energy Stent
Number analyzed (Participants) | 329
Percentage of participants | 99.4

13. Secondary Outcome: Lesion Success During the Index Procedure
Description: Evaluate the lesion success associated with the implant of the PRO-Kinetic Energy stent. Lesion success is defined as the successful delivery and deployment of the investigational stent at the intended target lesion in combination with any adjunctive device (if applicable) to attain a final residual stenosis of < 30% by operator visual estimate.
Time Frame: Index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Pro-Kinetic Energy Stent
Number analyzed (Participants) | 329
Percentage of participants | 99.4

14. Secondary Outcome: Angina Pectoris Classification
Description: Evaluate the angina pectoris classification at each study visit.
  Stable angina pectoris was classified according to the Canadian Cardiovascular Society's System: Stable Angina - Class I: normal activity does not cause angina; Stable Angina - Class II: slight limitation of normal activity, moderate exertion may cause angina; Stable Angina - Class III: marked limitation of ordinary physical activity; Stable Angina - Class IV: discomfort with any physical activity and pain may be present at rest
  Unstable angina pectoris was classified according to the Braunwald System: Numeral I: newly onset severe or accelerated angina with no pain at rest; Numeral II: angina at rest within the preceding month but not the past 48 hours Numeral III: angina at rest within the preceding 48 hours; Letter A: develops in presence of conditions which intensify ischemia; Letter B: develops in the absence of extracardiac conditions; Letter C: develops within 2 weeks after an acute myocardial infarction
Time Frame: Basline, Discharge, 1, 9, 12, 24 and 36 months post-index procedure
Population: Long term follow-up data collection is ongoing for the 12, 24 and 36 month intervals.
Measure: Number; unit: Percentage of participants
Groups:
- Pro-Kinetic Energy Stent - Baseline; PRO-Kinetic Energy Stent - Discharge; PRO-Kinetic Energy Stent - 1 Month; PRO-Kinetic Energy Stent - 9 Month; PRO-Kinetic Energy Stent - 12 Month; PRO-Kinetic Energy Stent - 24 Month; PRO-Kinetic Energy Stent - 36 Month: PRO-Kinetic Energy Stent: Coronary artery stent implant
Arm/Group | Pro-Kinetic Energy Stent - Baseline | PRO-Kinetic Energy Stent - Discharge | PRO-Kinetic Energy Stent - 1 Month | PRO-Kinetic Energy Stent - 9 Month | PRO-Kinetic Energy Stent - 12 Month | PRO-Kinetic Energy Stent - 24 Month | PRO-Kinetic Energy Stent - 36 Month
Number analyzed (Participants) | 329 | 329 | 326 | 307 | 303 | 296 | 283
Percentage of participants
  No Angina | 25.8 | 97.3 | 93.9 | 88.9 | 94.7 | 95.3 | 94.3
  Total Stable Angina | 61.7 | 2.4 | 5.8 | 11.1 | 5.0 | 4.7 | 4.9
  Stable Angina - Class I | 17.9 | 1.2 | 3.7 | 6.2 | 2.0 | 2.4 | 2.8
  Stable Angina - Class II | 23.4 | 0.6 | 0.9 | 2.9 | 1.7 | 1.0 | 1.4
  Stable Angina - Class III | 17.6 | 0.6 | 0.6 | 1.3 | 1.3 | 1.0 | 0.4
  Stable Angina - Class IV | 2.7 | 0.0 | 0.6 | 0.7 | 0.0 | 0.3 | 0.4
  Total Unstable Angina | 12.5 | 0.3 | 0.3 | 0.0 | 0.3 | 0.0 | 0.7
  Unstable Angine Class IA | 1.5 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Unstable Angine Class IB | 1.8 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Unstable Angine Class IC | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Unstable Angine Class IIA | 2.7 | 0.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Unstable Angine Class IIB | 2.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.7
  Unstable Angine Class IIC | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Unstable Angine Class IIIA | 1.2 | 0.0 | 0.0 | 0.0 | 0.3 | 0.0 | 0.0
  Unstable Angine Class IIIB | 3.0 | 0.0 | 0.3 | 0.0 | 0.0 | 0.0 | 0.0
  Unstable Angine Class IIIC | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: 36 Months
Arm/Group | Pro-Kinetic Energy Stent
All-Cause Mortality (participants affected / at risk) | 27/311
Serious Adverse Events (participants affected / at risk) | 202/329
Other Adverse Events (participants affected / at risk) | 118/329
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pro-Kinetic Energy Stent (N=329)
Atrial arrhythmia (Cardiac disorders) | 12 (13)
Ventricular arrhythmia (Cardiac disorders) | 3 (3)
Unspecified arrhythmia (Cardiac disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 4 (4)
Cardiac decompensation (Cardiac disorders) | 3 (6)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 3 (3)
Chest pain (Cardiac disorders) | 33 (42)
Congestive/worsening heart failure (Cardiac disorders) | 15 (16)
Diaphragmatic stimulation (Cardiac disorders) | 1 (1)
Dyspnea (Cardiac disorders) | 9 (9)
Edema (Cardiac disorders) | 3 (3)
Elective pacemaker/ICD implantation (Cardiac disorders) | 3 (3)
Elevated cardiac enzymes (Cardiac disorders) | 2 (2)
Heart block (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 6 (6)
Hypertensive urgency (Cardiac disorders) | 2 (2)
Ischemic cardiomyopathy (Cardiac disorders) | 1 (1)
Left ventricle penetration observed on LV gram (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 17 (20)
Palpitations (Cardiac disorders) | 3 (3)
Peri-procedural myocardial infarction (Cardiac disorders) | 1 (1)
Planned PCI procedure (Cardiac disorders) | 2 (2)
Planned routine angiography (Cardiac disorders) | 2 (2)
Pleural effusion (Cardiac disorders) | 4 (4)
Stenosis/occlusion of target lesion within non-study stented segment (Cardiac disorders) | 1 (1)
Stenosis/restenosis of non-target lesion in target vessel (Cardiac disorders) | 14 (19)
Stenosis/restenosis of non-target vessel (Cardiac disorders) | 27 (36)
Syncope (Cardiac disorders) | 3 (3)
Valvular heart disease (Cardiac disorders) | 5 (6)
Actinic keratosis/cheilitis (Skin and subcutaneous tissue disorders) | 1 (2)
Cicatricial changes to the left lower eyelid (Skin and subcutaneous tissue disorders) | 1 (1)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Non-healing wound (Skin and subcutaneous tissue disorders) | 1 (1)
Ulcer (Skin and subcutaneous tissue disorders) | 3 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia and/or hypomagnaesemia (Metabolism and nutrition disorders) | 3 (4)
Hypothyroidism (Endocrine disorders) | 1 (1)
Left adrenal mass (Endocrine disorders) | 1 (1)
Thyroid nodule (Endocrine disorders) | 1 (1)
Worsening diabetes (Endocrine disorders) | 2 (2)
Abdominal bloating (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Acute gangrenous cholecystitis (Gastrointestinal disorders) | 1 (1)
Anastomotic disruption (Gastrointestinal disorders) | 1 (1)
Atypical chest pain (Gastrointestinal disorders) | 1 (1)
Candida esophagitis (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Diverticulosis (Gastrointestinal disorders) | 2 (2)
Elective bariatric surgery (Gastrointestinal disorders) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 9 (10)
Gastritis (Gastrointestinal disorders) | 3 (3)
Heartburn (Gastrointestinal disorders) | 1 (1)
Intestinal ilius (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Nausea and/or vomiting (Gastrointestinal disorders) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 3 (4)
Septic shock (Gastrointestinal disorders) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Tubulovillous adenoma of ascending colon (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 7 (8)
Acute onset chronic renal injury (Renal and urinary disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 7 (7)
Contrast induced increased creatinine/acute renal insufficiency (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 4 (4)
Polyuria (Renal and urinary disorders) | 1 (1)
Prostatic bleeding (Renal and urinary disorders) | 1 (1)
Renal stone (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 10 (12)
Bleeding requiring treatment (Blood and lymphatic system disorders) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Coumadin toxicity (Blood and lymphatic system disorders) | 1 (1)
Hematoma - TAVI access site bleed (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (3)
Supratherapeutic INR (Blood and lymphatic system disorders) | 3 (4)
Bronchitis (Infections and infestations) | 7 (7)
Cellulitis (Infections and infestations) | 4 (4)
Fever (Infections and infestations) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
HSV pneumonitis (Infections and infestations) | 1 (1)
Leukocytosis (Infections and infestations) | 3 (3)
MRSA (Infections and infestations) | 2 (2)
Oral thrush (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 12 (17)
Sepsis (Infections and infestations) | 3 (4)
Surgical site dehiscence (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 11 (11)
Wound (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Calcar fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Genu varus deformity of right knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal injury/fall (Musculoskeletal and connective tissue disorders) | 11 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Vertebral fracture (Musculoskeletal and connective tissue disorders) | 2 (3)
Worsening/degenerative osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Encephalopathy (Nervous system disorders) | 6 (6)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Neuropathic pain (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 3 (4)
Transient ischemic attack (Nervous system disorders) | 3 (3)
Cataracts (Eye disorders) | 2 (2)
Eye irritation (Eye disorders) | 1 (1)
Herpes opthalmicus (Eye disorders) | 1 (1)
Low pupillary dilation (Eye disorders) | 1 (1)
Strabismus (Eye disorders) | 1 (1)
Depression with suicidal ideations (Psychiatric disorders) | 1 (1)
Major depression, chronic, recurrent with psychotic features (Psychiatric disorders) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 10 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
End-stage lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung rheumatism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Atypical chest pain (Cardiac disorders) | 4 (5)
Dehydration (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Extracardiac pain (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Steroid toxicogenic reaction (General disorders) | 1 (1)
Vasovagal episode (General disorders) | 1 (1)
Abdominal aortic aneurysm (Vascular disorders) | 3 (3)
Carotid artery disease (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Femoral artery thrombosis (Vascular disorders) | 1 (1)
Iliac artery stenosis / occlusion (Vascular disorders) | 2 (2)
Peripheral ischemia (Vascular disorders) | 9 (13)
Pseudoaneurysm (Vascular disorders) | 1 (1)
Systemic emboli - spleen (Vascular disorders) | 1 (1)
Vessel dissection or perforation (Vascular disorders) | 5 (5)
Worsening of peripheral artery disease (Vascular disorders) | 1 (1)
Worsening ulceration (Vascular disorders) | 1 (1)
Stenosis or occlusion of target lesion within stent segment (Vascular disorders) | 27 (33)
Stent thrombosis (Vascular disorders) | 5 (5)
Stent thrombosis, ARC assessment (Vascular disorders) | 9 (9)
Stent underexpansion (Vascular disorders) | 1 (1)
Vessel dissection or perforation during stenting procedure (Vascular disorders) | 8 (8)
Elevated troponin (Surgical and medical procedures) | 1 (1)
Hematoma (Surgical and medical procedures) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Relapsed myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cecum and liver cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Angina (Cardiac disorders) | 1 (2)
Arrhythmia, Ventricular Extrasystole (Cardiac disorders) | 1 (1)
Ascites (Cardiac disorders) | 1 (1)
Fatigue (Cardiac disorders) | 3 (3)
Hypotension (Cardiac disorders) | 3 (4)
Hypertrophic cardiomyopathy (Cardiac disorders) | 1 (1)
Non-specific ST-T changes (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Premature ventricular contractions (Cardiac disorders) | 1 (1)
Pulmonary hypertension (Cardiac disorders) | 1 (1)
Stenosis - location unknown (Cardiac disorders) | 1 (1)
Vasospasm (Cardiac disorders) | 1 (1)
Worsening Coronary Artery Disease (Cardiac disorders) | 3 (3)
Adrenal nodule (Endocrine disorders) | 1 (1)
Gout (Endocrine disorders) | 1 (1)
Hypoglycemia (Endocrine disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal incisional hernia (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gall bladder stone (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Hiatal hernie (Gastrointestinal disorders) | 1 (1)
Percutaneous endoscopic gastrostomy complication (Gastrointestinal disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Unbilica hernia (Gastrointestinal disorders) | 1 (1)
Benign prostatic hyperplasia (Renal and urinary disorders) | 1 (1)
Obstructive prostatism (Renal and urinary disorders) | 1 (1)
Hypovolemia (Blood and lymphatic system disorders) | 1 (1)
Subtherapeutic INR (Blood and lymphatic system disorders) | 1 (1)
Knee arthooplasty (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Pancreas infection (Infections and infestations) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left knee degenerative joint disease (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Right hand weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Ulnar fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Seisure (Nervous system disorders) | 1 (1)
spinal stenosis (Nervous system disorders) | 1 (1)
Syndope (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Acute renal injury (Renal and urinary disorders) | 2 (2)
Renal insufficiency (Renal and urinary disorders) | 1 (1)
Renal obstruction (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Fibrotic Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (2)
Peripheral vascular disease (Vascular disorders) | 1 (1)
Post-surgical bleeding (Vascular disorders) | 1 (1)
Saphenous vein insufficiency (Vascular disorders) | 1 (1)
Allergic reaction to contrast media (Immune system disorders) | 1 (1)
Allergic reaction with angioedema (Immune system disorders) | 1 (1)
Decreased hearing (Ear and labyrinth disorders) | 1 (1)
Dyspnea (General disorders) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Metabolic acidosis (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Syncope (General disorders) | 2 (2)
Possible PCI (Vascular disorders) | 1 (1)
Pacemaker manfunction (Cardiac disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pro-Kinetic Energy Stent (N=329)
Chest pain (Cardiac disorders) | 59 (77)
Dizziness (Cardiac disorders) | 31 (35)
Dyspnea (Cardiac disorders) | 44 (55)
Fatigue (Cardiac disorders) | 22 (30)
Hypertension (Cardiac disorders) | 30 (35)
Muskuloskeletal injury/fall (Cardiac disorders) | 18 (29)
Headache (General disorders) | 25 (30)
Atrial Arrhyrhmia (Cardiac disorders) | 17 (22)
Back Pain (Musculoskeletal and connective tissue disorders) | 18 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No